CLINICAL TRIAL: NCT07213687
Title: Effectiveness of Low-Dose Ketamine and Intravenous Lidocaine Versus Fentanyl for Postoperative Pain for Patients Undergoing Elective Gynecologic Surgery Under General Anesthesia: A Randomized Controlled Trial
Brief Title: Effectiveness of Low-Dose Ketamine and Intravenous Lidocaine Versus Fentanyl for Postoperative Pain
Acronym: Vs(versus)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dilla University (Other)
Responsible Party: Principal Investigator, Amanuel Asefa Akirso, Effectiveness of Low-Dose Ketamine and Intravenous Lidocaine Versus Fentanyl for Postoperative Pain for Patients Undergoing Elective Gynecologic Surgery, Dilla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: duirb/037/23-05
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: The eligible participants presenting for gynecologic surgery in both study areas will be allocated to study groups by a computer-generated random allocation sequence created by an independent anesthetist using Microsoft Excel 2016 with a 1:1 allocation to the treatment group (T) and control group (C). The treatment group will receive ketamine 0.5 mg/kg bolus, then 0.2 mg/kg infusion, and IV lidocaine 1.5 kg/kg bolus. The same bolus dose of lidocaine will be repeated every 15 to 20 minutes. The control group will receive a conventional GA with fentanyl 2µg/kg given during induction of anesthesia and one fourth of initial dose of fentanyl will be given over 20-30 minutes.
Who Masked: Participant
Masking Description: Only participants will not be allowed to now the group they allocated. The anesthetist involved in patient management will prepare drugs. Apart from patient management, the anaesthetist will not be involved in any other study processes. Participants will be given the study group code and allowed to present it to OR. Participants assigned to groups will not know which group they have been selected for.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- An Experimental or treatment group (T) (Experimental): The Experimental or treatment group (T) will receive ketamine 0.5 mg/kg bolus, then 0.2 mg/kg infusion, and IV lidocaine 1.5 kg/kg bolus. The same bolus dose of lidocaine will be repeated every 15 to 20 minutes.
  Interventions: Drug: Low dose intravenous ketamine
- Control group (C) (Active Comparator): The control group (C) will receive a conventional general anesthesia (GA) with fentanyl 2µg/kg given during induction of anesthesia and one fourth of initial dose of fentanyl will be given over 20-30 minutes.
  Interventions: Drug: Low dose intravenous ketamine

INTERVENTIONS:
Drug: Low dose intravenous ketamine — Patients in the treatment group will be administered through a Ketamine IV bolus of 0.5 mg/kg during the induction phase with propofol of 3 mg/kg, followed by a continuous infusion of ketamine of 0.2 mg/kg/hr. Before induction, a lidocaine bolus of 1.5 mg/kg will be given, and the same dose of lidocaine will be administered every 15 to 20 minutes after induction of anesthesia until the start of skin closure. Patients in control group will receive a conventional GA with fentanyl 2µg/kg given during induction of anesthesia and one fourth of initial dose of fentanyl will be given over 20-30 minutes.
  Other Names: Intravenous lidocaine; Intravenous fentanyl

SUMMARY:
Background: Rational approaches to perioperative patient management have been used to meet intraoperative analgesic needs and avoid opioid-related adverse effects. A combination of drugs, such as ketamine, sodium channel blockers, anti-inflammatories, and alpha-2 agonists, can be used. This study aimed to compare the effectiveness of low-dose ketamine and intravenous lidocaine with fentanyl for intraoperative pain in patients undergoing gynecologic surgery.

Objective: To determine the effectiveness of low-dose ketamine and intravenous lidocaine versus fentanyl for postoperative pain in patients undergoing elective gynecologic surgery under general anesthesia at Dilla University General and Teaching Hospital from April 10, 2023, to June 10, 2023.

Methodology: A randomized, controlled, single-blind trial will be conducted with 68 adult patients undergoing elective gynecologic surgery under GA. Eligible patients undergoing gynecologic surgery in both study areas will be allocated by a computer-generated random allocation sequence in equal ratios to the treatment group (T) receiving low-dose ketamine and IV lidocaine and the control group (C) receiving fentanyl. The primary outcome variable is the postoperative pain score measured at PACU, 6 hours, 12 hours, and 24 hours postoperatively. Secondary outcomes are analgesic consumption, postoperative hypoxemia, Quality of immediate postoperative recovery assessed by the quality of recovery (QoR-40) questionnaire on postoperative days 1, and postoperative nausea and vomiting. It will be collected up to 24 hours postoperatively. Data will be analyzed using Student's t-test, analysis of variance, chi-square test, and Mann-Whitney test. Parametric and non-parametric categorical data will be analyzed using the chi-squared test and Fisher's exact test, respectively. Statistical significance will be a p-value of 0.05.

Work plan and budgeting: - study will be conducted from April 10, 2023, to June 10, 2023, with a cost of 41625 ETB.

DETAILED DESCRIPTION:
After obtaining ethical clearance from Dilla University College of Health Sciences and Medicine's ethics review board, a structured questionnaire will be developed and translated into the respective languages by the principal investigator (PI). Two BSC anesthetists involved in patient management will be selected at the study area and trained in the overall process of participant handling and data collection.

During the preoperative period Patients undergoing gynecologic operations during the study period will be assessed and informed about the study process and anesthesia on the day before surgery. The patient will receive maintenance fluid, have bilateral peripheral IV lines secured, and will be NPO the night before surgery. On the morning of the procedure, both a standard informed consent form for the procedure and a separate consent form for the study were available.

The availability and functionality of the bilateral IV line and NPO status will be checked, and prophylactic drugs will be given. Standard preoperative questionnaires were used, and data were collected through patient responses and medical records, such as patient monitoring and charts.

During the intraoperative period Routine ASA monitoring will be checked and applied for patients in both groups when they present to the OR. The functionality and availability of the bilateral IV line and urinary catheter were rechecked. Propofol (3 mg/kg) was used to induce anesthesia after the patient had been pre-oxygenated for both groups. An intravenous bolus of 0.5 mg/kg of ketamine during the induction phase for patients in the treatment group, then a continuous infusion of 0.2 mg/kg/hr. 0f ketamine. A bolus of 1.5 mg/kg was given before induction, and the same dose of lidocaine was administered every 15 to 20 minutes after induction of anesthesia until the start of skin closure.

Patients in the control group were induced with fentanyl 2 μg/kg given during induction of anesthesia with propofol 3mg/kg. 0.5 μg /kg of fentanyl was given every 20-30 minutes up to the start of skin closure.

Intubation was performed after giving 1.5-2 mg/kg IV suxamethonium. Inhalational anesthetics as availabilities (Isoflurane 0.75-2% and Halothane 1%_ 2%) were opened after the position of the ETT was confirmed, and Dexamethasone 0.15mg/kg IV bolus was given after securing the ETT.

Anesthesia was maintained with inhalational agents according to the patient's tidal volume of 6-8 ml/kg adjusted to maintain oxygen saturation >95% with 3- 4 ml 100% oxygen flow, and end-tidal CO2 between 32 and 45 mmHg. Muscle relaxation was maintained with vecuronium 0.8 mg/kg. Intraoperative anesthesia depth was assessed by clinical signs as well as by patient monitoring. Estimated intraoperative blood loss was supplied with ringer lactate or normal saline.

The intraoperative participants' data were collected from the anesthesia record chart and patient monitoring. Intraoperative hemodynamic variables were collected every 10 minutes. Intraoperative cardiac adverse events such as intraoperative bradycardia (pulse rate less than 50 bpm), tachycardia (PR greater than 100 bpm), hypertension, and hypotension we diagnosed and managed as per institutional protocol. Intraoperative nausea or vomiting in both groups was also managed as an institutional protocol.

When the surgeon began skin closure, the inhalational agent turned off. A pre-prepared reversal agent bolus (neostigmine 0.05 mg/kg with atropine 0.02 mg/kg IV) was administered for patients given long-acting muscle relaxants after checking the adequacy of spontaneous ventilation, adequate movement of the respiratory bag, oxygen saturation >95percentage and ETCO2 between 32 and 45 mmHg after the skin is closed.

During the postoperative period The postoperative pain severity was assessed by the validated VAS starting from the patient's discharge from PACU to 24 hours postoperatively. Data was collected at discharge from PACU, at 6 hours, 12 hours, and 24 hours postoperatively. PONV data were collected from the time of arrival at PACU at 6 hours, 12 hours, and 24 hours postoperatively according to the patient's signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients between the ages of 18 and 65 undergoing elective gynecologic surgery under general anaesthesia

Exclusion Criteria:

* Patients with allergies to any of the drugs used in the trial Patients with chronic pain Patients who are diagnosed with CNS diseases like psychiatric diseases, epilepsy Patients who are hypertensive and taking beta blockers, as well as those who have preoperative bradycardia, hypotension, or any type of heart block, Breastfeeding and pregnant women Patients weighing less than 40 kg or obese patients (BMI > 35 kg/m2) Patients with a history of smoking

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult patients between the ages of 18 and 65 will undergo elective gynecologic surgery under general anesthesia
Enrollment: 70 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
The numerical rating scale will measure the postoperative pain severity | From the patient's arrival at PACU to 24 hours postoperatively (at PACU, at 6 hours, 12 hours, and 24 hours).
  Will be assessed by the validated numerical rating scale, a reliable tool for assessing pain intensity in all populations, regardless of literacy level which employs a 0-to-10 ratings. scale, with 0 representing no pain and 10 representing the worst possible pain. The English and Amharic versions of the scale are attached in

SECONDARY OUTCOMES:
The occurrence of postoperative nausea and vomiting (PONV) | At arrival at PACU to 24hours (at PACU, at 6 hours, 12 hours, and 24 hours)
  The occurrence of postoperative nausea and vomiting, the nausea and vomiting score, and the use of medication for management will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Amanuel A Asefa, Msc. Degree, Principal Investigator — Arbaminch College of Health Sciences
Locations (1):
- Dilla University, Awasa, Snnpr, Ethiopia

IPD SHARING:
Plan to Share IPD: No
will share after the final result.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT07213687/Prot_SAP_ICF_000.pdf